CLINICAL TRIAL: NCT05662670
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of WJ13405 Monotherapy in Patients With Advanced or Mentastatic Non-Small Cell Lung Cancer
Brief Title: A Phase I/II Study of WJ13404 Monotherapy in Patients With Advanced or Mentastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the adjustment of the R&D strategy, Suzhou Junjing Biosciences Co., Ltd. decided to terminate this study in September 2023
Sponsor: Suzhou Junjing BioSciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS113-001-I
Record Dates: First submitted 2022-11-11; First posted 2022-12-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:WJ13404 tablets (Experimental): Dose escalation: 6 dose levels The dose escalation study is proposed to include 6 dose levels: 30, 90, 180, 270, 360, and 480 mg once daily.
  (It can be adjusted based on clinical PK data and safety results after discussion between PI and the sponsor).
  Dose-expansion: After the initial data evaluation, the Sponsor and the SMC will select 2-3 dose levels to evaluate drug safety and PK further, explore its preliminary efficacy, and determine RP2D.
  Efficacy expansion: The RP2D determined in dose escalation and dose expansion will be applied.
  Interventions: Drug: WJ13404 tablets

INTERVENTIONS:
Drug: WJ13404 tablets — Dose escalation: 6 dose levels The dose escalation study is proposed to include 6 dose levels: 30, 90, 180, 270, 360, and 480 mg once daily.
  (It can be adjusted based on clinical PK data and safety results after discussion between PI and the sponsor).
  Dose-expansion: After the initial data evaluation, the Sponsor and the SMC will select 2-3 dose levels to evaluate drug safety and PK further, explore its preliminary efficacy, and determine RP2D.
  Efficacy expansion: The RP2D determined in dose escalation and dose expansion will be applied.

SUMMARY:
This is an open-label phase I/II preliminary study, including dose escalation, dose expansion, and efficacy expansion, to evaluate drug safety, tolerability, PK, and efficacy. The dose escalation study evaluates the IMP's safety, tolerability, and PK in patients with locally advanced or metastatic NSCLC who have experienced disease progression after third-generation EGFR-TKI therapy. The dose expansion study, after 2-3 dose levels are selected based on dose escalation results, further investigates the IMP's safety, tolerability, and PK, explores preliminary efficacy, and determines RP2D in patients with locally advanced or metastatic NSCLC harboring EGFR C797X mutation. The efficacy expansion study evaluates the IMP's safety and efficacy in patients with locally advanced or metastatic NSCLC harboring EGFR C797X mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old, male or female;
2. Histologically or cytologically confirmed locally advanced or recurrent/metastatic advanced NSCLC that is inoperable, is subject to progression or intolerability after the standard of care, or is unable to be treated or has not been treated by the standard of care;
3. Dose escalation: patients with EGFR sensitive mutation who have experienced disease progression after third-generation EGFR-TKI therapy;
4. Dose expansion and efficacy expansion: patients with proven EGFR C797X mutation;
5. Patients who agree to provide tumor tissues and blood samples for EGFR mutation analysis (certain patients who are unable to provide qualified tumor tissues may be enrolled once approved by investigators and the Sponsor);
6. At least one measurable lesion as per RECIST v1.1;
7. ECOG PS score of 0-1;
8. Expected survival of more than 12 weeks;
9. Sufficient vital organ functions at screening (requiring no blood transfusion, use of hematopoietic stimulating factor, or use of human albumin preparation within 14 days before screening):

   1. ANC ≥ 1.5 × 109/L;
   2. Platelet ≥ 100 × 109/L;
   3. Hemoglobin > 90 g/L;
   4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.0 × upper limit of normal (ULN) (in the presence of liver metastasis, ≤ 5 × ULN);
   5. Total bilirubin (TBIL) ≤ 1.5 × ULN;
   6. Coagulation function (INR) ≤ 1.5 × ULN;
   7. Blood creatinine ≤ 1.5 × ULN or creatinine clearance (Ccr, calculated by the Cockcroft-Gault formula) ≥ 45 mL/min;
   8. Serum lipase and amylase ≤ 1.5 × ULN;
10. Females with childbearing potential and a negative serum pregnancy test within 7 days before enrollment who agree to use effective contraception during the IMP treatment and 6 months after the last dose. This protocol defines "females with childbearing potential" as sexually mature women who: 1) have not undergone a hysterectomy or bilateral ovariectomy; 2) have not had spontaneous menopause for 24 consecutive months (i.e., no menstrual bleeding at any time within the last 24 consecutive months; amenorrhea after cancer treatment does not indicate infertility). Male patients whose sexual partners are females with childbearing potential must agree to use effective contraception during the study treatment and 6 months after the last dose;
11. Patients who voluntarily participate in this study and have signed the informed consent form after an all-inclusive informed consent process.

Exclusion Criteria:

1. Patients who have received systemic anti-tumor therapy within 4 weeks before the first dose, including chemotherapy, targeted therapy, anti-vascular drug therapy, biologic therapy, immunotherapy, radiotherapy, or other IMP therapy; moreover, patients who have received EGFR-TKI targeted therapy may be enrolled if 5 half-lives have passed after discontinuation;
2. Patients who are receiving strong CYP3A inhibitors or inducers; or those who have yet to reach 5 half-lives after discontinuation of a strong inhibitor, or 5 half-lives or 14 days (whichever is longer) after discontinuation of a strong inducer at the time of the first WJ13404 dosing;
3. Patients who have experienced adverse events caused by previous anti-tumor therapy that have yet to improve to CTCAE v5.0 grade ≤ 1 at screening (except for neurotoxicity and alopecia, which cannot be recovered as assessed by investigators);
4. Patients who are plagued by other malignancies (except for non-melanoma basal or squamous cell carcinoma of the skin, carcinoma in situ of the breast/cervix, superficial bladder cancer, thyroid cancer, and other carcinomas in situ, treated with curative intent and without evidence of recurrent disease) concurrently or within 5 years before treatment initiation;
5. History of diseases causing chronic diarrhea, including but not limited to Crohn's disease and irritable bowel syndrome;
6. Active gastrointestinal disease or other conditions that may significantly compromise drug absorption, metabolism, or excretion;
7. Patients known to have undergone organ transplantation or stem cell transplantation; patients who have undergone major surgery or serious trauma within 4 weeks before the first dose (excluding needle biopsy for sample collection);
8. Patients who are suffering from carcinomatous meningitis and spinal cord compression;
9. Patients who meet one of the following cardiac criteria: Unexplained or cardiovascular-caused presyncope or syncope, ventricular tachycardia, ventricular fibrillation, or cardiac arrest, with average corrected QT interval (based on 3 ECGs taken at rest, QTc, using the Fridericia's correction formula) > 450 ms in males or > 470 ms in females. Various clinically significant cardiac rhythm, conduction, or resting ECG morphological abnormalities, such as complete left bundle branch block, third-degree conduction block, second-degree conduction block, PR interval > 250 ms, and echocardiography-suggested left ventricular ejection fraction (LVEF) < 50%. Various factors that may increase the risks of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, history of immediate family members with long QT syndrome or sudden death of unknown cause before age 40, and current receipt of any drug known to prolong the QT interval;
10. Unstable systemic diseases, such as active infection requiring systemic drug therapy, poorly controlled hypertension, unstable angina, congestive heart failure, serious hepatic, renal, or metabolic conditions including cirrhosis, renal failure, and uremia;
11. Patients who experience dyspnea or require continuous oxygen therapy, or who are suffering from CTCAE v5.0 grade ≥ 2 active pneumonitis or interstitial lung disease (except mild radiation pneumonitis);
12. Central nervous system metastasis with symptoms. Patients who have received treatment for brain metastases may be considered for enrollment, provided that no disease progression confirmed by radiologic imaging evaluation occurs within 4 weeks before the first dose of the IMP, no evidence shows new or enlarging brain metastases, and radiation, surgery, or steroid therapy has been discontinued for at least 4 weeks before the first dose of the IMP;
13. HBV-RNA > upper limit of the reference value when positive for hepatitis B surface antigen or hepatitis B core antibody;
14. HCV-RNA > upper limit of the reference value when positive for hepatitis C antibody;
15. Positive for human immunodeficiency virus (HIV);
16. Patients with a confirmed history of mental disorders who are receiving drugs for treatment;
17. History of substance or drug abuse;
18. Patients who have received traditional Chinese medicine for anti-tumor therapy within 1 week before the first dose of the study treatment;
19. Previous serious eye disorders that have not recovered to grade ≤ 1;
20. Skin toxicity at > grade 2 within 4 weeks before the first dose;
21. Pregnancy and lactation;
22. Other factors, as evaluated by investigators, that have potential effects on study results and may interfere with the patient's participation, including previous or existing physical conditions (such as eye disorders, including corneal ulcers and conjunctivitis), treatment or laboratory test abnormalities, patient unwillingness to abide by the study procedures, restrictions, and requirements, and the presence of psychological or social conditions that may interfere with their participation or affect the study result evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
adverse events（AE) and serious adverse events（SAE) | up to 3 years
  To evaluate incidence，severity and outcome of adverse events（AE),and serious adverse events（SAE)
ORR | up to 3 years
  Proportion of patients who have the best response of confirmed or partial response as per RECIST v1.1.ORR, along with its 95% CI, will be calculated
DLT | up to 2 years (only for dose escalation and dose expansion）
  DLT is defined as any of the following toxicities that occur during the DLT observation and are deemed by investigators possibly, probably, or definitely related to WJ13404 as per NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Cmax | up to 3 years
  It's suitable for dose escaltion and does extension ,maximum plasmaconcentration
Tmax | up to 3 years
  It's suitable for dose escaltion and does extension,time to Cmax
AUC 0-t | up to 3 years
  It's suitable for dose escaltion and does extension,area under the concentration versus time curve from time 0 to the last measurable concentration.
t1/2 | up to 3 years
  It's suitable for dose escaltion and does extension, elimination half-life.
CL/F | up to 3 years
  It's suitable for dose escaltion and does extension, clearance.
Vd/F | up to 3 years
  It's suitable for dose escaltion and does extensionapparent volume of distribution
λz | up to 3 years
  It's suitable for dose escaltion and does extension, elimination rate constant.
Css-min | up to 3 years
  It's suitable for dose escaltion and does extension,minimum concentration at steady state.
Css-max | up to 3 years
  It's suitable for dose escaltion and does extension,maximum concentration at steady state.
Css-ave | up to 3 years
  It's suitable for dose escaltion and does extension, average concentration at steady state.
AUCtau-ss | up to 3 years
  It's suitable for dose escaltion and does extension,area under the concentration versus time curve for a dosing interval at steady state.
Vss | up to 3 years
  It's suitable for dose escaltion and does extension,volume of distribution at steady state.
AR | up to 3 years
  It's suitable for dose escaltion and does extension,accumulation ratio.
DF | up to 3 years
  It's suitable for dose escaltion and does extension,degree of fluctuation.
ORR | up to 3 years
  It's suitable for dose escaltion and does extension, objective response rate.
DOR | up to 3 years
  It's suitable for dose escaltion and does extension, duration of response.
DCR | up to 3 years
  It's suitable for dose escaltion and does extension, disease control rate.
PFS | up to 3 years
  It's suitable for dose escaltion and does extension, progression-free survival.
OS | up to 3 years
  It's suitable for dose escaltion and does extension,overall survival.
adverse events（AE) and serious adverse events（SAE) | up to 1 years（only for efficacy expansion stage）
  To evaluate incidence，severity and outcome of adverse events（AE),and serious adverse events（SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided